CLINICAL TRIAL: NCT00005452
Title: Ti PC Software for Analyzing Longitudinal Data
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4385; R44HL047237 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To develop TI (pronounced 'T-sub-I'), a personal computer program to analyze time-varying data generated by periodic patient reports, repeatedly-observed disease signs, or serial biomarkers to study chronic disease.

DETAILED DESCRIPTION:
BACKGROUND:

With the advent of quasi-likelihood, generalized estimating equations, and new ways to handle missing data, has come a striking increase in applicable models, perhaps more than after the 1972 introduction of the Cox model for survival data. TI provided a way to analyze the data.

DESIGN NARRATIVE:

TIl provided graphics for data exploration and model validation. TI ran under most current version of Windows, used Civilized Software's MLAB as its programming language, offered context-sensitive help, a dictionary of relevant terms, identification of file entries from their screen position, and simple animation. TI permitted the user to analyze time-varying data from the two perspectives of repeated measured using a variety of models and time series where both time and frequency domain tools were provided.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-09; Study Completion 1996-04 (Actual)